CLINICAL TRIAL: NCT06819293
Title: A Phase I, Open Label, Single Center Study Evaluating the Safety and Efficacy of IB-T101 Injection for Treatment of Patients with Advanced Clear Cell Renal Cell Carcinoma
Brief Title: IB-T101 Injection for Treatment of Patients with Advanced Clear Cell Renal Cell Carcinoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Grit Biotechnology (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GTE-002-001
Record Dates: First submitted 2025-02-05; First posted 2025-02-11 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Advanced Clear Renal Cell Carcinoma; Adult

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- IB-T101 injection treatment group (Experimental)
  Interventions: Biological: IB-T101 injection

INTERVENTIONS:
Biological: IB-T101 injection — IB-T101 injection to treat advanced clear renal cell carcinoma

SUMMARY:
This is an open label, single center, dose escalation, and dose extension IIT study aimed at evaluating the safety, efficacy, and pharmacokinetics of IB-T101 in adult patients with advanced clear renal cell carcinoma

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily join the study, signed informed consent form， willing and able to comply with the study protocol;
2. Age ≥18 years old;
3. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1;
4. Expected survival time of ≥ 3 months;

Exclusion Criteria:

1. CNS dysfunction with clinical significance. For example, seizures, cerebral ischemia/hemorrhage, dementia, cerebellar diseases, cerebral edema, reversible posterior encephalopathy syndrome, or any autoimmune disease involving the CNS.
2. Any form of primary and acquired immunodeficiency (such as severe combined immunodeficiency). Known human immunodeficiency virus (HIV) positive subjects
3. Have experienced myocardial infarction or unstable angina within the 6 months prior to screening
4. Pleural effusion requiring drainage for symptom management within 28 days prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-12-06 (Actual); Primary Completion 2027-12-07 (Estimated); Study Completion 2027-12-07 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 3 years
  To evaluate efficacy parameters such Objective Response Rate(ORR) per RECIST v1.1, as assessed by the Investigater
AEs | 3 years
  To characterize thesafty profile of autologous TIL injection IB-T101 in patients with advanced fclear renal cell carcinoma as measured by the incidence and severity of adverse events per CTCAE 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji hospital, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No